CLINICAL TRIAL: NCT06562504
Title: Transcranial Electrical Stimulation Combined With Interim Testing Promotes Temporal Memory in Patients With Schizophrenia
Brief Title: Temporal Memory in Schizophrenic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaofeng Ma (Other)
Responsible Party: Sponsor-Investigator, Xiaofeng Ma, Professor, Northeast Normal University
Organization: Northeast Normal University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: No.2024018
Record Dates: First submitted 2024-08-15; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Patients With Schizophrenia
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anodal group (Experimental): In the anodal group, the anode was placed over the left DLPFC (F3), and the cathode was placed over the contralateral supraorbital area (FP2). A direct current of 2mA was applied for 20 minutes during each stimulation session.
  Interventions: Device: Transcranial direct current stimulation (tDCS)- anodal group
- Sham group (Sham Comparator): In the sham group, the stimulation parameters, including the stimulation site and duration, were identical to those of the anodal group. However, during the 10-second ramp-up and ramp-down periods before and after stimulation, patients were unaware that the current was turned off.
  Interventions: Device: Transcranial direct current stimulation (tDCS)- sham group
- tACS group (Experimental): In the transcranial alternating current stimulation (tACS) group, the anode was placed in the left DLPFC (F3) and the cathode was placed in the contralateral supraorbital region (FP2). A direct current of 1.5 mA was applied for 20 minutes during each stimulation, theta rhythm, 6 HZ.
  Interventions: Device: transcranial alternating current stimulation (tACS)-tACS group

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS)- anodal group — 2mA/20mins/session;
  Arms: Anodal group
Device: Transcranial direct current stimulation (tDCS)- sham group — 0mA/20mins/session
  Arms: Sham group
Device: transcranial alternating current stimulation (tACS)-tACS group — 1.5 mA/20 min/session; 6HZ, theta
  Arms: tACS group

SUMMARY:
Temporal order memory deficits are a central feature of cognitive abnormalities in schizophrenia. The dorsolateral prefrontal cortex contributes to the extraction of temporal contextual information. Transcranial direct current stimulation (tDCS) and interim testing have been shown to be external techniques that can improve temporal order memory deficits in schizophrenia patients. Transcranial alternating current stimulation (tACS) can also improve cognitive functioning in patients with schizophrenia. This study intends to investigate the learning effects of temporal order memory under two learning strategies during tDCS targeting the left dorsolateral prefrontal cortex (L-DLPFC) and transcranial direct current stimulation (tDCS) interventions in patients with schizophrenia, to investigate whether it can promote the retention of temporal order memory in patients, and to compare the differences in the effects of the two intervention modalities.

This study was planned to recruit 75 patients diagnosed with schizophrenia from the hospital.

A single online tDCS (2 mA × 20 min) and tACS (1.5 mA × 20 min, theta rhythm) intervention was conducted during which participants performed a temporal-sequence memory task for visual pictures, and test scores were compared for each stimulus type on an intermediate test and repetition of the two strategies of learning.

DETAILED DESCRIPTION:
Treatment was conducted by two examiners, and participants' memory levels were tested before the start of the experiment using a flanker task and a numerical breadth task as baseline tests. The experimental procedure was divided into a learning phase, in which participants memorized the sequence of pictures, and a testing phase, in which participants were required to recall a picture presented after the probe item. Participants were randomly assigned in parallel to each stimulus type and learning strategy, with 25 receiving tdcs anodized stimuli, 25 receiving sham stimuli, and another 25 receiving tacs stimuli. And participants' inhibitory control continued to be tested using the flanker task before and after the stimuli for pre- and post-intervention comparisons.

ELIGIBILITY:
Inclusion Criteria:

1. Meeting the diagnostic criteria for schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5);
2. Aged 18 years or older, regardless of gender, with an educational level of elementary school or above;
3. All patients received stable-level antipsychotic medication treatment, were in a stable phase of disease treatment, able to understand the testing requirements, and cooperated to complete all research tasks;
4. No history of neurological disorders or other serious physical illnesses, and no history of intellectual disability;
5. No color blindness, color weakness, or other color vision impairments, with normal vision or corrected vision.

Exclusion Criteria:

1. Clear cognitive impairment caused by somatic or cerebral organic lesions, such as cerebrovascular diseases, traumatic brain injury, etc;
2. Individuals with mental disorders caused by substance dependence or abuse, or the use of psychoactive substances;
3. History of brain injury or other central nervous system-related organic diseases;
4. Individuals at significant risk of suicide or harming others;
5. Participation in similar experiments in the past 30 days prior to baseline.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Correctness of temporal recall | 5mins to 24 hours
  Stimulus content was presented using the Eprime experimental program, and participants pressed key responses during the test phase to record their rate of correctness.
  Stimulus content was presented using the Eprime experimental program, and participants pressed key responses during the test phase to record their rate of correctness.
proactive interference rate | 5mins to 24 hours
  The rate of intrusion of prior information when participants recalled the current information was counted.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Ma, Professor, Principal Investigator — Northwest Normal University
Locations (1):
- Northwest Normal University, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2024-07-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT06562504/Prot_000.pdf
  • Informed Consent Form (2024-07-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT06562504/ICF_001.pdf